CLINICAL TRIAL: NCT00710437
Title: Effects of Dexmedetomidine on the Intraoperative Electroencephalogram During Endarterectomy Surgery
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200513433; 200513433-1 (Other: UC Davis, Institutional Review Board); 200513433-2 (Other: UC Davis, Institutional Review Board); 200513433-3 (Other: UC Davis, Institutional Review Board); 200513433-4 (Other: UC Davis, Institutional Review Board); 200513433-5 (Other: UC Davis, Institutional Review Board)
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Endarterectomy, Carotid
Keywords: Dexmedetomidine; Carotid Endarterectomy; Electroencephalogram
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Dexmedetomidine - used
  Interventions: Drug: Dexmedetomidine
- 2: Dexmedetomidine - not used
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Steady state infusion 0.007 mcg/kg/min

SUMMARY:
During elective carotid endarterectomy surgery, dexmedetomidine, an FDA approved medication, is now given as part of our standard anesthetic regimen based upon its reported ability to decrease anesthetic requirements and improve the peri-operative hemodynamic profile without compromising the EEG monitoring that is used during these procedures. Although this is consistent with our clinical impression, the effects of dexmedetomidine on the perioperative course and EEG monitoring have not been objectively evaluated at our institution.

DETAILED DESCRIPTION:
Fifty sequential patient records will be identified from a search of the OR surgical schedules and reviewed: 25 patients before the introduction of dexmedetomidine and a standard anesthetic protocol and 25 patients after the introduction of the protocol. Data will be collected during an individual review of the pre-operative anesthetic evaluation, the intra-operative anesthetic record and the post-anesthesia care unit record and collated in an Excel spread sheet kept on a secure personal computer in the PI's office. All personal identifiers will be removed and the patients numbered sequentially before and after introduction of the clinical protocol. The data collected will be used to characterize the intraoperative anesthetic requirements, effects on EEG activity and the immediate postoperative recovery period. The review is expected to require 2 months to complete.

This review will be restricted to records that already exist. No therapeutically removed tissues will be collected. There will be no additional tests. No blood samples will be collected. No additional procedures are involved in this study activity. There is no incomplete disclosure.

The resources and personnel are currently available to complete this review. The entire project including data collection, analysis and summarization will be completed by the PI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective carotid endarterectomy

Exclusion Criteria:

* Emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2005-04; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Effects of Dexmedetomidine on the Intraoperative Electroencephalogram During Endarterectomy Surgery | April 2005 - November 2009
  Data collection and analysis complete. Permanently closed.

CONTACTS AND LOCATIONS:
Overall Officials: Neal W Fleming, M.D., Ph.D., Study Director — Director, Cardiovascular and Thoracic Anesthesiology, UC Davis, Department of Anesthesiology and Pain Medicine
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States